CLINICAL TRIAL: NCT02601287
Title: A Safety and Efficacy Study of Botulinum Toxin Type A (BOTOX®) to Treat Urinary Incontinence Due to Neurogenic Detrusor Overactivity or Overactive Bladder in Korean Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191622-151
Record Dates: First submitted 2015-11-06; First posted 2015-11-10 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOTOX® 100U (Experimental): Botulinum Toxin Type A 100U into the detrusor muscle on Day 1 in patients with Overactive Bladder
  Interventions: Biological: Botulinum Toxin Type A
- BOTOX® 200U (Experimental): Botulinum Toxin Type A 200U into the detrusor muscle on Day 1 in patients with Neurogenic Detrusor Overactivity
  Interventions: Biological: Botulinum Toxin Type A

INTERVENTIONS:
Biological: Botulinum Toxin Type A — Botulinum Toxin Type A into detrusor muscle on Day 1
  Other Names: BOTOX®; onabotulinumtoxinA

SUMMARY:
This is a safety and efficacy study of BOTOX® (Botulinum Toxin Type A) in the Treatment of Adult Korean Patients with Urinary Incontinence due to Neurogenic Detrusor Overactivity or Overactive Bladder.

ELIGIBILITY:
Inclusion Criteria:

* Urinary incontinence as a result of neurogenic overactive bladder due to spinal cord injury or multiple sclerosis
* Symptoms of urge urinary incontinence, urgency, and frequency due to overactive bladder

Exclusion Criteria:

* Myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
* Use of botulinum toxin therapy of any serotype in the 3 months prior to screening
* Has acute urinary retention who do not routinely perform clean intermittent self-catheterization (CIC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from the baseline in the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) total score | Baseline, Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Medical Contact, Study Director — Allergan
Locations (5):
- South Korea (5):
  - Pusan National University Hospital, Busan, Korea
  - The Catholic University of Korea Bucheion St. Mary Hospital, Gyeonggi-do, Korea
  - Seoul National University Hospital, Seoul, Korea
  - Asan Medical Center, Seoul, Korea
  - Samsung Medical Center, Seoul, Korea